CLINICAL TRIAL: NCT02116894
Title: Phase Ib Study of the Combination Regorafenib With PF-03446962 in Patients With Refractory Metastatic Colorectal Cancer (REGAL-1 Trial)
Brief Title: Safety Study of Regorafenib With PF-03446962 to Treat Colorectal Cancer
Acronym: REGAL-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jeffrey Clarke, Principal Investigator, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00051541
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; PF-03446962; regorafenib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ascrinvacumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PF-03446962 plus regorafenib (Experimental)
  Interventions: Biological: PF-03446962; Drug: Regorafenib

INTERVENTIONS:
Biological: PF-03446962 — PF-03446962 will be an investigational formulation supplied by Pfizer . PF-03446962 injection, 10 mg/mL is presented as a sterile solution for IV administration in a formulation consisting of precedented excipients. We will be administering PF-03446962 intravenously at a starting dose of 4.5 mg/kg and escalating to up to 7 mg/kg.
Drug: Regorafenib — We will be administering regorafenib on-label for the indication of metastatic colorectal cancer. The indicated dose is 160 mg once daily for the first 21 days of a 28 day cycle. We will start at a regorafenib dose of 120 mg in the combination therapy, but may increase to 160 mg during dose escalation.

SUMMARY:
The primary objective of this open-label phase Ib trial is to determine the maximum tolerated dose and the recommended phase II dose for the combination of PF-03446962 plus regorafenib in patients with metastatic colorectal cancer. The secondary objectives are to describe the safety and tolerablility, and to describe the clinical activity of PF-03446962 plus regorafenib in terms of response rate and progression free survival

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed and radiographically evaluable refractory metastatic colorectal adenocarcinoma for which regorafenib would be considered a therapeutic option.
2. Disease must be measurable by RECIST 1.1 criteria (see Appendix 1).
3. Age ≥ 18 years.
4. ECOG 0 or 1.
5. Life expectancy of at least 3 months.
6. Adequate bone marrow function as shown by:

   1. ANC ≥ 1.5 x 109
   2. Platelets ≥ 100 x 109/L
   3. Hemoglobin ≥ 9 g/dL; Erythropoietin and transfusion support is permitted provided treatments are not required more than every 8 weeks. Hemoglobin must be stable above or equal to 9 g/dL for at least 2 weeks prior to day 1of study drug without blood transfusion to maintain hemoglobin level.
7. Adequate liver function as shown by:

   1. serum bilirubin ≤ 1.5x ULN
   2. PT/PTT/INR ≤ 1.5x ULN
   3. ALT and AST ≤ 2.5x ULN
8. Adequate renal function: creatinine clearance (estimated) ≥ 50 cc/min by Cockroft Gault or 24 hour urine (see Appendix 6).
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days from day 1 of study drug; both men and women must be willing to use two methods of contraception, one of them being a barrier method during the study and for 6 months after last study drug administration.
10. Signed informed consent.
11. Presence of an archived tumor sample (no size requirements).

Exclusion Criteria:

1. Prior regorafenib use with disease progression (expanded cohort only).
2. Prior failure to tolerate regorafenib at 120 mg/day.
3. Patients currently receiving anticancer therapies or who have received anticancer therapies within 28 days from day 1 of study drug (including investigational agents, chemotherapy, radiation therapy, antibody based therapy, etc.)
4. Patients who:

   1. Have had a major surgery or significant traumatic injury within 4 weeks from day 1 of study drug,
   2. Have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or
   3. Are anticipated to require major surgery during the course of the study.
5. Patients who have exhibited hypersensitivity reactions to regorafenib and/or a structural compound, biological agent, or formulation (eg sorafenib).
6. Grade 3-4 AE associated with prior anti-VEGF therapy. Grade 3 hypertension that was readily managed will be permitted.
7. History of grade 3 or higher hypersensitivity reactions/anaphylaxis attributed to humanized and/or chimeric monoclonal antibodies or other such proteins. Hypersensitivity reactions that are clearly related to cetuximab may be permitted at the discretion of the principal investigator.
8. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent with the following exceptions:

   1. Intermittent steroids (not to exceed 4 mg every day) may be used on an as-needed basis (e.g. treatment for chemotherapy-related nausea, anorexia and fatigue.)
   2. Patients on physiologic replacement doses of steroids due to adrenal insufficiency for any reason may remain on these medications.
   3. Topical, inhaled or intra-articular corticosteroids
9. Active brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Treated, asymptomatic metastases are permitted provided the patient has been off steroids for at least 1 month prior to day 1 of study drug.
10. Severe chronic obstructive or other pulmonary disease with hypoxemia (requires supplementary oxygen, symptoms due to hypoxemia or O2 saturation <90% by pulse oximetry after a 2 minute walk or in the opinion of the investigator any physiological state likely to cause systemic or regional hypoxemia.
11. Presence of poorly controlled atrial fibrillation (ventricular heart rate >100 bpm)
12. Previous history of CVA, TIA, angina pectoris, acute MI or history of recent re-perfusion procedures (e.g. PTCA), pulmonary embolus or untreated deep vein thrombosis (DVT) within 6 months from day 1 of study drug. NOTE: Subjects with recent DVT who have been therapeutically anti-coagulated for at least 6 weeks are eligible.
13. Known significant or active CAD or PVD or CVD defined as abnormal stress test, symptoms, or requiring medication for the prevention of symptoms.
14. Congestive heart failure (New York Heart Association (NYHA classification, see Appendix 4 functional classification III-IV).
15. Proteinuria at screening demonstrated by urine analysis (UA) > 1+ and 24 hour urine protein ≥ 1 gram/24 hours.
16. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study as so judged by the treating physician. Examples include but are not limited to:

    1. Severely impaired lung function (e.g. use of home O2, history of Idiopathic Lung Disease (ILD), any evidence of ILD on scan.
    2. Active (acute or chronic) severe infections requiring treatment with I.V. antibiotics.
    3. Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
    4. Poorly controlled hypertension [defined as systolic blood pressure (SBP of >140 mmHg or diastolic blood pressure (DBP) of >90 mmHg] NOTE: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. Following antihypertensive medication initiation or adjustment, blood pressure (BP) must be re-assessed three times at approximately 2-minute intervals. At least 24 hours must have elapsed between anti-hypertensive medication initiation or adjustment and BP measurement. These three values should be averaged to obtain the mean diastolic blood pressure and the mean systolic blood pressure. The mean SBP/DBP ratio must be <140/90 mmHg in order for a subject to be eligible for the study.
17. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral medications (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
18. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to day 1 of study drug
19. History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) or other significant spontaneous bleeding event within 1 month prior to day 1 of study drug or at any time on a prior VEGF inhibitor.
20. History of abdominal fistula or gastrointestinal perforation at any point within 6 months prior to day 1 of study drug, unless surgically repaired.
21. Active peptic ulcer disease, inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation or gastrointestinal bleeding.
22. Use or need for full dose anticoagulation other than low molecular weight heparin and Factor Xa inhibitors (e.g. Lovenox, Fondaparinux) and no other bleeding risk.
23. Serious, non-healing wound, active ulcer, or untreated bone fracture as judged by treating physician.
24. Active bleeding diathesis.
25. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
26. Known history of HIV or Hepatitis B or C seropositivity.
27. Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Two acceptable forms of contraceptives must be continued throughout the trial by either sex and for 2 months (60 days) following last dose of either drug. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to day 1 of study drug).
28. Concomitant use of CYP3A4 strong inducers and strong inhibitors. (See Appendix 7).
29. Corrected QTc interval > 500 msec. If QTc interval is > 500 msec, then 2 additional ECGs should be obtained over a brief period of time (e.g., within 15-20 minutes) to confirm the abnormality. The average QTc interval will be determined from the 3 ECG tracings by manual evaluation and will be used to determine if the subject will be excluded from the study. The same method of QTc determination must be used throughout the subject's participation in the trial.
30. History of Osler-Weber-Rendu syndrome or Hereditary Hemorrhagic Telangiectasia
31. Patients unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RPTD) for the combination of PF-03446962 plus regorafenib | RPTD for the study will be determined at the completion of Phase I dose escalation cohort; estimated as 1 year

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of PF 03446962 administered in combination with regorafenib | Continuous, every 4 weeks minimum until end of study estimated at 4 years
  Adverse events will be recorded
Response rate of PF 03446962 plus regorafenib | approximately every 8 weeks and/or restaging
  Response is assessed at restaging, approximately every 8 weeks, assessed for an average of 6 months
Progression free survival associated with PF 03446962 plus with regorafenib | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Duke University Medical Center, Durham, North Carolina, United States